CLINICAL TRIAL: NCT03840005
Title: A Phase II, Placebo Controlled, Double Blind, Randomised Clinical Trial To Assess The Safety And Tolerability Of 30mg/kg Daily Ursodeoxycholic Acid (UDCA) In Patients With Parkinson's Disease (PD)
Brief Title: Trial of Ursodeoxycholic Acid (UDCA) for Parkinson's Disease: The "UP" Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: JP Moulton Charitable Foundation (Other); PRO.MED.CS Praha a.s. (Unknown); Clinical Trials Research Unit, University of Sheffield (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STH18493; 2018-001887-46 (EudraCT Number)
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A randomised double-blind, placebo controlled 48 week trial of UDCA at a daily dose of 30 mg/kg in patients with early Parkinson's disease <3 years post diagnosis.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind trial. The investigators, clinical study team, participants and analysing statistician will be blind to treatment allocation. The active treatment will be over-encapsulated and a matched placebo manufactured to maintain the blind.
  The Independent Data Monitoring Committee (IDMC) is the only oversight body that has access to unblinded accumulating comparative data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 2:1 in favour of UDCA
  Interventions: Drug: Ursonorm
- Ursonorm (Ursodeoxycholic acid) (Experimental): UDCA 30 mg/kg daily, tablet form taking orally , administered 3 monthly for 12 months, dose titration during the 1st month will occur.
  Interventions: Drug: Ursonorm

INTERVENTIONS:
Drug: Ursonorm — Ursodeoxycholic acid
  Other Names: UDCA

SUMMARY:
The aim of this study is to explore the potential of Ursodeoxycholic acid (UDCA) to slow down the progression of Parkinson's Disease (PD) in a randomised, double-blind, placebo-controlled, "proof of concept" study. The primary objective of the study will be to determine the safety and tolerability of this drug in patients with PD. Participants will be recruited form a cohort of patients who have been diagnosed with PD within the last 3 years and are potentially suitable for this study.

There is strong evidence from previous research and the work carried out by other groups that UDCA rescues the function of the mitochondria (mitochondria are the "powerhouse" of the cell) in PD patient tissue and other models of PD. This suggests that UDCA may slow down the worsening of PD.

UDCA has been in clinical use for the treatment of liver disease (primary biliary cholangitis) for over 30 years. The investigators therefore know that it is safe and well tolerated in patients with liver disease but the investigators don't know yet whether this is also the case in patients with PD. Furthermore, the dose used for patients with liver disease (15 mg/kg) is not high enough for UDCA to get into the brain. The investigators therefore need to double the dose to 30 mg/kg. This higher dose was also safe in clinical trials for liver disease, but is currently not used routinely in clinical practice.

DETAILED DESCRIPTION:
The primary aim of this study is to generate clinical data to examine the safety, tolerability & potential effectiveness of 48 weeks exposure to UDCA compared to placebo. Furthermore, it will determine the usefulness of novel objective readouts (namely the objective sensor based quantification of motor progression & 31P-MRS/imaging-based in vivo quantification of ATP) which may allow a reduction of the sample size (& thus cost) of future trials.

This is double-blind, randomised, placebo-controlled multi-centre parallel group trial in patients with PD who have been diagnosed ≤ 3 years ago. 30 patients will be randomised to UDCA at a dose of 30 mg/kg or matched placebo using a 2:1 split (20 patients on UDCA, 10 on placebo). This will include 48 week exposure period & a subsequent 8 week washout period. Detailed evaluations of all patients will take place at Screening, Baseline, 12, 24, 36, 48 & 56 weeks. The trial medication will be taken at 3 equal doses per day, to be taken orally with food. The dose will be increased gradually by 250 mg (1 capsule) every 3 days until patient reaches a dose of 30 mg/kg.

Visit Schedule

Telephone Contact 1 (Telephone Screening)

Subsequent to the site staff having received a reply slip from the patient indicating their interest to participate in the study, a suitable time & date will be arranged with the respective patient to undergo telephone screening by a member of the research team to check potential eligibility, including a brief review of relevant medical history. The Chief Investigator (CI)/ Principal Investigator (PI) will check the screening record made after the telephone screening call. Any patients not deemed eligible to be invited for their screening visit will be contacted by a member of the research team to inform them of this outcome. Patients deemed eligible will be invited to a screening visit. The date of diagnosis & confirmation of the PD diagnosis & any other uncertainties relating to the inclusion/exclusion criteria will be confirmed subsequent to this telephone screening assessment for those patients who seem eligible but are outside the Sheffield Teaching Hospitals (STH)/ University College London Hospitals (UCLH) geographical area by requesting copies of relevant clinic letters or contacting their PD Clinical Consultants directly. The telephone screening call will be repeated if the patient cannot attend visit 0 (screening visit) within 1-8 weeks to ensure that s/he would still fulfil the telephone screening eligibility criteria.

The telephone screening call will not be undertaken for study patients who are already patients of either site.

Visit 0: Screening (Time -1 - 8 weeks prior to baseline visit)

At this visit the research team will answer any further questions, check the patient's eligibility for the study as far as possible and, if the patient wishes to participate in the study, obtain written consent. A clinical diagnosis of PD is based on the opinion of the Principal Investigator (PI) after review of the patient's clinical history, examination findings & response to PD medication.

The written informed consent process will be undertaken by the PI or by an appropriately trained member of the research team as delegated by the PI/ CI. This study will not include vulnerable patients or patients who lack capacity.

Screening procedures

The PI (or authorised delegate) will complete the following screening assessments/procedures with the patient:

* Obtaining consent
* Inclusion/Exclusion Review
* Demographic information & medical history
* Demographic data regarding PD
* Past medical history
* Medication History
* Family history
* Previous imaging
* Previous genetic tests
* Confirmation of eligibility
* Confirmation of date for diagnosis of Parkinson's disease by PIs or other experts in movement disorders (this may include review of medical records)
* Concomitant medication
* Physical examination (including assessment of modified Hoehn & Yahr stage), including weight, height &vital signs
* Montreal Cognitive Assessment (MoCA)
* Montgomery-Asberg Depression rating scale (MADRS)
* Confirmation of post-menopausal state
* Safety bloods (full blood count, urea & electrolytes, liver function tests, blood glucose, HbA1C, lipid profile)
* Serum sample (approach. 20 ml stored at -80 degrees Celsius)
* ECG
* Provision of physical activity monitor & activity diary

Assuming that the patient fulfils the immediate eligibility criteria, arrangements will be made for the patient to attend a baseline appointment approximately 2 to 4 weeks after the screening visit. This interval enables review of the patient's blood results to confirm final eligibility. If more than 8 weeks have elapsed since the screening visit, the screening visit & screening assessments should be repeated before proceeding to the baseline visit.

Patients who consent to the study but who are subsequently found not to meet the study eligibility criteria will be contacted by the research nurse or other member of the research team to inform them that they are not eligible to join the study. If any concerns about the patient's health or well-being are identified from out-of-range blood results or abnormal assessment scores, a member of the research team will inform the patient's General Practitioner (GP).

Following written consent, randomisation will take place at the baseline visit. All patients will be assigned a unique patient ID number at screening that will link all of the clinical information collected for them on the study database, these will be in the format Sxx/nnnn; where xx is a unique number assigned to the site by the Trial Manager & nnnn is a unique number starting at 0001 &incrementing by 1. Once the patient ID number has been entered, the system will supply a randomisation number which will identify the treatment pack to be dispensed. The randomisation will be 2:1 in favour of UDCA. The randomization system will stratify by site.

Site Study Teams

The local PI, supported by an appropriate member of the research team will monitor patient well-being, record adverse events, titrate &prescribe study medication. Since the 'treating' nurse or doctor will review all blood results & be aware of any reported side effects, a separate member of the research team will act as a blinded assessor, undertaking the MDS-UPDRS & other outcome measures after appropriate training. Ideally the blinded assessor will undertake the MDS-UPDRS Part 3 with the patient in the "OFF" state, followed by the complete MDS-UPDRS, Non-Motor Symptom assessment Scale (NMS-Quest) & MADRS once the patient is in the "ON" state. The practically defined "OFF" medication state refers to the patient assessment conducted in the absence of their regular medication with the aim of exposing the severity of the underlying PD. Efforts should be made to ensure that the same outcome assessor is present at all visits but sites should identify back-up personnel to cover staff absences & avoid cross-over of 'assessing' &'treating' team members.

Baseline (Visit 1)

Eligible patients will attend a further clinic visit where baseline assessments will be performed. Results of blood tests & ECG will be reviewed prior to baseline evaluation to ensure patient eligibility. They will be asked to attend in the "practically defined OFF" state. The following assessment will be undertaken in the "practically defined OFF" state:

* Confirmation of eligibility/inclusion/exclusion review
* Medication review
* Physical examination
* Recording of any Adverse Events (AEs)
* MDS-UPDRS part 3 (motor examination)
* Optogait &Opals sensor-based objective quantification of motor impairment (Sheffield Patients only)

They will be invited to take their PD medication following the assessment. The PI or authorised delegate will record any reported serious adverse events & changes to concomitant medications, including PD medication. In addition, the predicted progression will be calculated, following the model developed by Williams-Gray & co-workers. The Prognostic Model developed by Williams-Gray &co-workers identified the following three parameters as associated with more rapid PD progression: 1. Higher age, 2. Higher UPDRS motor examination axial score (items 27-30), 3. Lower animal naming fluency (patients will be asked to name as many animals as possible in a 1-minute time frame). The assessor will then complete the following procedures with the patient in the "practically defined ON" stage (typically 30-60 min after patient has taken PD symptomatic medication):

* MDS-UPDRS
* NMS-Quest
* PDQ-39
* 31P- MRS
* Blood sample for genetic analysis
* Safety bloods
* Serum sample
* Provision of patient diary
* Return of physical activity monitor &activity diary

Patients will be randomised at this visit to receive either active of placebo medication (2:1 ratio). The PI or appropriately delegated medically qualified member of the study team will complete &sign a study-specific prescription form for presentation to pharmacy by the patient. The prescription form will details the baseline medication allocation print-out from the randomisation computer system.

All patients will be provided with a study-specific diary by their local research team at the baseline visit, in which to record any alterations in the dose of trial medication or concomitant medications taken. Patients should be advised to contact the study team promptly should they develop loose stools rather than waiting for the next study visit or scheduled telephone call.

Visit 2: 12 week follow-up clinic

Patients will attend a clinic visit twelve weeks after the baseline visit, having taken all medications as usual. The PI or authorised delegate will complete the following procedures with the patient in conjunction with study diary review:

* Record any AEs & changes to concomitant medications
* Assess compliance with study treatment & collect any unused medication
* Return of unused medication
* Safety bloods
* Serum sample
* Diary Review

Provided that there are no immediate clinical contra-indications, the patient will be provided with a further 3 months prescription for the trial medication.

Visit 3: 24 week follow-up clinic

Patients will attend a clinic visit six months after the baseline visit, having taken all medications as usual. The PI or authorised delegate will complete the following procedures with the patient in conjunction with study diary review:

* Record any AEs & changes to concomitant medications
* ECG
* Safety bloods
* Serum sample
* Assess compliance with study treatment & collect any unused medication
* Return of unused medication
* MDS-UPDRS/part 3 motor assessment in the practically defined "ON" stage
* Diary Review

Provided that there are no immediate clinical contra-indications, the patient will be provided with a further 3 months prescription for the trial medication.

Visit 4: 36 week follow-up clinic

Patients will attend a clinic visit thirty six weeks after the baseline visit, having taken all medications as usual. The PI or authorised delegate will complete the following procedures with the patient in conjunction with study diary review:

* Record any AEs & changes to concomitant medications
* Assess compliance with study treatment & collect any unused medication
* Return of unused medication
* Safety bloods
* Serum sample
* Diary Review

Provided that there are no immediate clinical contra-indications, the patient will be provided with a further 3 months prescription for the trial medication.

Visit 5: 48 week follow-up clinic

Patients will attend a clinic visit 48 weeks after the baseline visit. For this visit, patients will be asked to attend on the day of assessment in the 'practically-defined OFF' state.

The assessor will complete the following procedures with the patients in conjunction with study diary review:

* Record any AEs & changes to concomitant medications
* Assess compliance with study treatment & collect any unused medication
* MDS-UPDRS part 3 in the "practically defined OFF" state
* Opticals/Sensor based gait assessment (Sheffield patients only)
* Height & Weight

Patients will then be invited to take their routine PD medication. The assessor will then complete the following procedures with the patient in the "practically-defined ON" state (typically 30 - 60 min later):

* MDS-UPDRS
* NMS-Quest
* MoCA
* MADRS
* PDQ-39
* Safety bloods
* Serum sample stored
* 31P- MRS
* Diary review
* Return of the physical activity monitor &activity diary

Visit 6: 56 week follow-up clinic

Patients will attend a clinic visit 56 weeks after the baseline visit. For this visit, patients will be asked to attend on the day of assessment in the 'practically-defined OFF' state. The PI or authorised delegate will complete the following procedures with the patient:

* Record any AEs & changes to concomitant medications
* Safety bloods
* Serum sample
* MDS-UPDRS part 3 motor subscale in the "practically defined OFF medication state"

Patients will then be invited to take their routine PD medication. The assessor will then complete the following procedures with the patient in the "practically-defined ON" state" (typically 30 - 60 min later):

* MDS-UPDRS
* NMS-Quest
* MoCA
* MADRS
* PDQ-39
* Diary review
* Diary collection

For all visits, each procedure is undertaken as part of the study & not part of the patient's standard care.

Telephone contacts There will be 12 telephone contacts throughout the study, weekly after the baseline visit during the dose escalation period &week 8, week 18, week 30, week 42 & week 52. Patients will also be contacted via the telephone 2 days prior to their baseline visit, visit 5 & visit 6 to remind patients to attend their next visit in the "practically defined OFF medication state" for their next visit.

Sensors At the screening visit, eligible patients will be given the DynaPort Movemonitor to wear for 7 days. A text message will be sent to the patients every morning to remind them to wear the device. A 2nd DynaPort Movemonitor will be posted to patients 2 weeks prior to their 48 week visit with instructions to wear the sensor for 7 days prior to their next visit. Patients will then be asked to return this at their 48 week visit.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosis of Parkinson's disease: PD is a clinical diagnosis as defined by the Queen Square Brain Bank criteria (bradykinesia defined as slowness of initiation of voluntary movement with progressive reduction in speed and amplitude on repetitive actions and at least one of the following: Rigidity, 4-6 Hz rest tremor). The diagnosis will have been made by the treating clinician and confirmed by the PI on site after review of the clinical history, examination findings and response to PD medication.

The Queen Square brain bank criteria MAY be used to help assist in the diagnosis although this need not be a formal inclusion criteria, and the relevance of a positive family history of PD, or a confirmed genetic basis for an individual's symptoms will be evaluated in the context of other clinical features in determining diagnosis and eligibility.

* Diagnosis of Parkinson's disease ≤ 3 years ago by a clinician with particular expertise in the diagnosis and treatment of movement disorders (typically one of the PIs or their consultant colleagues). The date of diagnosis will be verified by a review of the medical records.
* Subjective improvement of motor impairment on dopaminergic medication, confirmed by PI through personal examination and/or review of medical records
* Hoehn and Yahr stage ≤ 2.5 in the practically defined "ON" medication state. This implies that all patients will be mobile without assistance during their best "ON" medication periods.
* Ability to take study drug
* Ability to communicate in English
* Age 18 - 75 yr of any gender
* Documented informed consent to participate
* Able to comply with study protocol and willing to attend necessary study visits

Exclusion Criteria:

* Diagnosis or suspicion of other cause of parkinsonism such as Multiple system atrophy (MSA) or progressive supranuclear palsy (PSP), drug induced parkinsonism, dystonic tremor or essential tremor will not be recruited.
* Known abnormality on CT or MRI brain imaging considered likely to compromise compliance with trial/protocol/31P-MRS acquisition.
* Known claustrophobia or other reasons why patient could not tolerate or be suitable for 31P-MR Spectroscopy (31P-MRS)
* Current or previous exposure to UDCA
* Current or previous diagnosis of liver disease judged to be significant by the clinical investigator, in particular Primary Biliary Cholangitis (previously referred to as Primary Biliary Cirrhosis, PBC)
* Prior intracerebral surgical intervention for PD (including deep-brain stimulation). Patients who have previously undergone deep brain stimulation, intracerebral administration of growth factors, gene therapies or cell therapies will not be eligible.
* Already actively participating in a trial of a device, drug or surgical treatment for PD
* History of alcoholism
* Women of child - bearing potential (WOCBP)
* Participants who lack the capacity to give informed consent
* Any medical or psychiatric condition which in the investigator's opinion compromises the potential participant's ability to participate
* Concurrent dementia defined by Montreal Cognitive assessment (MoCA) score <25
* Concurrent severe depression defined by a score >16 on the Montgomery- Asberg Depression Rating Scale (MADRS)
* Serum transaminases (such as aspartate transaminase (AST) more than 2 times upper limit of normal.
* Patients on ciclosporin, nitrendipine or dapsone for the treatment of concomitant, general medical conditions.
* Participants with previous or current diagnosis of inflammatory bowel disease (i.e. ulcerative colitis or Crohn's disease)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Incidence of Treatment-Emergent Adverse Events | Timepoint: start of treatment to 56 weeks (visit 6)
  Safety of a 56-week UDCA Intervention will be assessed by measuring the number of participants with adverse events that are related to treatment.
Number of Participants with Incidence of Serious Adverse Events | Timepoint: start of treatment to 56 weeks (visit 6)
  Safety of a 56-week UDCA Intervention will be assessed by measuring the number of participants with serious adverse events.
Number of Participants that complete the study | Timepoint: start of treatment to 56 weeks (visit 6)
  Safety of a 56-week UDCA Intervention will be assessed by measuring the number of participants that complete the study.

SECONDARY OUTCOMES:
Mean change from baseline to week 48 in participant scores on the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part 3 motor subsection in the "OFF" medication state. | Timepoint: 48 weeks (visit 5)
  Motor symptoms will be measured using the MDS-UPDRS part 3 motor subsection. Part III of the scale will be completed at baseline, visit 3 (24 weeks), visit 5 (48 weeks).
  The scale consists of four parts; Part I "Non-motor experiences of daily living" (13 questions), Part II "Motor Experiences of daily living" (13), Part III "Motor Examination" (33) and Part IV "Motor Complications" (6). Each question has five responses that are linked to common clinical terms: 0=Normal, 1=Slight, 2=Mild, 3=Moderate, 4=Severe. Whereas each response is tailored to the question, the progression of impairment is based on consistent infrastructure. "Slight" refers to symptoms with sufficiently low frequency/intensity to cause no impact on function; "Mild" refers to symptoms of frequency/intensity sufficient to cause modest impact on function; "Moderate" refers to symptoms sufficiently frequent/intense to impact considerably, but not prevent, function; "Severe" refers to symptoms that prevent function.
Mean change from baseline to week 48 in in vivo parameter estimates of Adenosine Triphosphate (ATP) levels, derived from participant cranial 31P-Magnetic Resonance Spectroscopy (MRS) centered on the basal ganglia and related motor regions. | Timepoint: 48 weeks (visit 5)
  Patients who consent to having the 31P-MR spectroscopy, data will be analysed for the change in energy metabolic levels at baseline and visit 5 (week 48).
Mean change from baseline to week 48 in in vivo parameter estimates of Phosphocreatinine (PCr) levels, derived from participant cranial 31P-Magnetic Resonance Spectroscopy (MRS) centered on the basal ganglia and related motor regions. | Timepoint: 48 weeks (visit 5)
  Patients who consent to having the 31P-MR spectroscopy, data will be analysed for the change in energy metabolic levels at baseline and visit 5 (week 48).
Mean change from baseline to week 48 in in vivo parameter estimates of Inorganic Phosphate (Pi) levels , derived from participant cranial 31P-Magnetic Resonance Spectroscopy (MRS) centered on the basal ganglia and related motor regions. | Timepoint: 48 weeks (visit 5)
  Patients who consent to having the 31P-MR spectroscopy, data will be analysed for the change in energy metabolic levels at baseline and visit 5 (week 48).
Mean change from baseline to week 48 in objective quantification of participant motor impairment, using motion sensors. | Timepoint: 48 weeks (visit 5)
  For the subset of patients who consent to having the Opticals sensor based gait assessment, the data will be analysed for changes in motor impairment at baseline and visit 5 (week 48).

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Bandmann, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire
  - University College London Institute of Neurology, London

IPD SHARING:
Plan to Share IPD: Yes
The results of this trial will be submitted for publication in a peer reviewed journal, in addition to reports at appropriate specialist conferences. The results of the trial will be disseminated regardless of the direction of effect. No participants will be identified during this process.
Supporting Information: Study Protocol
Time Frame: Requests for the supporting information will be considered on a case by case basis with the CI and sponsor in conjunction with contract agreements with collaborators
Access Criteria: As above

REFERENCES:
- [Background] Velseboer DC, de Bie RM, Wieske L, Evans JR, Mason SL, Foltynie T, Schmand B, de Haan RJ, Post B, Barker RA, Williams-Gray CH. Development and external validation of a prognostic model in newly diagnosed Parkinson disease. Neurology. 2016 Mar 15;86(11):986-93. doi: 10.1212/WNL.0000000000002437. Epub 2016 Feb 17. PMID 26888991
- [Background] Kalia LV, Lang AE. Parkinson's disease. Lancet. 2015 Aug 29;386(9996):896-912. doi: 10.1016/S0140-6736(14)61393-3. Epub 2015 Apr 19. PMID 25904081
- [Background] Findley LJ, Wood E, Lowin J, Roeder C, Bergman A, Schifflers M. The economic burden of advanced Parkinson's disease: an analysis of a UK patient dataset. J Med Econ. 2011;14(1):130-9. doi: 10.3111/13696998.2010.551164. PMID 21235405
- [Background] Kordower JH, Olanow CW, Dodiya HB, Chu Y, Beach TG, Adler CH, Halliday GM, Bartus RT. Disease duration and the integrity of the nigrostriatal system in Parkinson's disease. Brain. 2013 Aug;136(Pt 8):2419-31. doi: 10.1093/brain/awt192. PMID 23884810
- [Background] Schapira AH, Olanow CW, Greenamyre JT, Bezard E. Slowing of neurodegeneration in Parkinson's disease and Huntington's disease: future therapeutic perspectives. Lancet. 2014 Aug 9;384(9942):545-55. doi: 10.1016/S0140-6736(14)61010-2. Epub 2014 Jun 18. PMID 24954676
- [Background] Exner N, Lutz AK, Haass C, Winklhofer KF. Mitochondrial dysfunction in Parkinson's disease: molecular mechanisms and pathophysiological consequences. EMBO J. 2012 Jun 26;31(14):3038-62. doi: 10.1038/emboj.2012.170. PMID 22735187
- [Background] Gasser T. Usefulness of Genetic Testing in PD and PD Trials: A Balanced Review. J Parkinsons Dis. 2015;5(2):209-15. doi: 10.3233/JPD-140507. PMID 25624421
- [Background] Auburger G, Klinkenberg M, Drost J, Marcus K, Morales-Gordo B, Kunz WS, Brandt U, Broccoli V, Reichmann H, Gispert S, Jendrach M. Primary skin fibroblasts as a model of Parkinson's disease. Mol Neurobiol. 2012 Aug;46(1):20-7. doi: 10.1007/s12035-012-8245-1. Epub 2012 Feb 19. PMID 22350618
- [Background] Mortiboys H, Johansen KK, Aasly JO, Bandmann O. Mitochondrial impairment in patients with Parkinson disease with the G2019S mutation in LRRK2. Neurology. 2010 Nov 30;75(22):2017-20. doi: 10.1212/WNL.0b013e3181ff9685. PMID 21115957
- [Background] Mortiboys H, Thomas KJ, Koopman WJ, Klaffke S, Abou-Sleiman P, Olpin S, Wood NW, Willems PH, Smeitink JA, Cookson MR, Bandmann O. Mitochondrial function and morphology are impaired in parkin-mutant fibroblasts. Ann Neurol. 2008 Nov;64(5):555-65. doi: 10.1002/ana.21492. PMID 19067348
- [Background] Mortiboys H, Furmston R, Bronstad G, Aasly J, Elliott C, Bandmann O. UDCA exerts beneficial effect on mitochondrial dysfunction in LRRK2(G2019S) carriers and in vivo. Neurology. 2015 Sep 8;85(10):846-52. doi: 10.1212/WNL.0000000000001905. Epub 2015 Aug 7. PMID 26253449
- [Background] Mortiboys H, Aasly J, Bandmann O. Ursocholanic acid rescues mitochondrial function in common forms of familial Parkinson's disease. Brain. 2013 Oct;136(Pt 10):3038-50. doi: 10.1093/brain/awt224. Epub 2013 Sep 2. PMID 24000005
- [Background] Chun HS, Low WC. Ursodeoxycholic acid suppresses mitochondria-dependent programmed cell death induced by sodium nitroprusside in SH-SY5Y cells. Toxicology. 2012 Feb 26;292(2-3):105-12. doi: 10.1016/j.tox.2011.11.020. Epub 2011 Dec 8. PMID 22178905
- [Background] Greene LA, Levy O, Malagelada C. Akt as a victim, villain and potential hero in Parkinson's disease pathophysiology and treatment. Cell Mol Neurobiol. 2011 Oct;31(7):969-78. doi: 10.1007/s10571-011-9671-8. Epub 2011 Mar 10. PMID 21547489
- [Background] Abdelkader NF, Safar MM, Salem HA. Ursodeoxycholic Acid Ameliorates Apoptotic Cascade in the Rotenone Model of Parkinson's Disease: Modulation of Mitochondrial Perturbations. Mol Neurobiol. 2016 Mar;53(2):810-817. doi: 10.1007/s12035-014-9043-8. Epub 2014 Dec 15. PMID 25502462
- [Background] Castro-Caldas M, Carvalho AN, Rodrigues E, Henderson CJ, Wolf CR, Rodrigues CM, Gama MJ. Tauroursodeoxycholic acid prevents MPTP-induced dopaminergic cell death in a mouse model of Parkinson's disease. Mol Neurobiol. 2012 Oct;46(2):475-86. doi: 10.1007/s12035-012-8295-4. Epub 2012 Jul 8. PMID 22773138
- [Background] Ward A, Brogden RN, Heel RC, Speight TM, Avery GS. Ursodeoxycholic acid: a review of its pharmacological properties and therapeutic efficacy. Drugs. 1984 Feb;27(2):95-131. doi: 10.2165/00003495-198427020-00001. PMID 6365507
- [Background] Crosignani A, Setchell KD, Invernizzi P, Larghi A, Rodrigues CM, Podda M. Clinical pharmacokinetics of therapeutic bile acids. Clin Pharmacokinet. 1996 May;30(5):333-58. doi: 10.2165/00003088-199630050-00002. PMID 8743334
- [Background] Abbas G, Lindor KD. Pharmacological treatment of biliary cirrhosis with ursodeoxycholic acid. Expert Opin Pharmacother. 2010 Feb;11(3):387-92. doi: 10.1517/14656560903493460. PMID 20102304
- [Background] Parry GJ, Rodrigues CM, Aranha MM, Hilbert SJ, Davey C, Kelkar P, Low WC, Steer CJ. Safety, tolerability, and cerebrospinal fluid penetration of ursodeoxycholic Acid in patients with amyotrophic lateral sclerosis. Clin Neuropharmacol. 2010 Jan-Feb;33(1):17-21. doi: 10.1097/WNF.0b013e3181c47569. PMID 19935406
- [Background] Carey EJ, Ali AH, Lindor KD. Primary biliary cirrhosis. Lancet. 2015 Oct 17;386(10003):1565-75. doi: 10.1016/S0140-6736(15)00154-3. Epub 2015 Sep 11. PMID 26364546
- [Background] Siegel JL, Jorgensen R, Angulo P, Lindor KD. Treatment with ursodeoxycholic acid is associated with weight gain in patients with primary biliary cirrhosis. J Clin Gastroenterol. 2003 Aug;37(2):183-5. doi: 10.1097/00004836-200308000-00018. PMID 12869893
- [Background] Ratziu V, de Ledinghen V, Oberti F, Mathurin P, Wartelle-Bladou C, Renou C, Sogni P, Maynard M, Larrey D, Serfaty L, Bonnefont-Rousselot D, Bastard JP, Riviere M, Spenard J; FRESGUN. A randomized controlled trial of high-dose ursodesoxycholic acid for nonalcoholic steatohepatitis. J Hepatol. 2011 May;54(5):1011-9. doi: 10.1016/j.jhep.2010.08.030. Epub 2010 Oct 31. PMID 21145828
- [Background] Cullen SN, Rust C, Fleming K, Edwards C, Beuers U, Chapman RW. High dose ursodeoxycholic acid for the treatment of primary sclerosing cholangitis is safe and effective. J Hepatol. 2008 May;48(5):792-800. doi: 10.1016/j.jhep.2007.12.023. Epub 2008 Feb 14. PMID 18314215
- [Background] Angulo P, Dickson ER, Therneau TM, Jorgensen RA, Smith C, DeSotel CK, Lange SM, Anderson ML, Mahoney DW, Lindor KD. Comparison of three doses of ursodeoxycholic acid in the treatment of primary biliary cirrhosis: a randomized trial. J Hepatol. 1999 May;30(5):830-5. doi: 10.1016/s0168-8278(99)80136-6. PMID 10365809
- [Background] Shineman DW, Alam J, Anderson M, Black SE, Carman AJ, Cummings JL, Dacks PA, Dudley JT, Frail DE, Green A, Lane RF, Lappin D, Simuni T, Stefanacci RG, Sherer T, Fillit HM. Overcoming obstacles to repurposing for neurodegenerative disease. Ann Clin Transl Neurol. 2014 Jul;1(7):512-8. doi: 10.1002/acn3.76. Epub 2014 Jun 24. PMID 25356422
- [Background] Ackerman HD, Gerhard GS. Bile Acids in Neurodegenerative Disorders. Front Aging Neurosci. 2016 Nov 22;8:263. doi: 10.3389/fnagi.2016.00263. eCollection 2016. PMID 27920719
- [Background] Olanow CW, Schapira AH, LeWitt PA, Kieburtz K, Sauer D, Olivieri G, Pohlmann H, Hubble J. TCH346 as a neuroprotective drug in Parkinson's disease: a double-blind, randomised, controlled trial. Lancet Neurol. 2006 Dec;5(12):1013-20. doi: 10.1016/S1474-4422(06)70602-0. PMID 17110281
- [Background] Athauda D, Maclagan K, Skene SS, Bajwa-Joseph M, Letchford D, Chowdhury K, Hibbert S, Budnik N, Zampedri L, Dickson J, Li Y, Aviles-Olmos I, Warner TT, Limousin P, Lees AJ, Greig NH, Tebbs S, Foltynie T. Exenatide once weekly versus placebo in Parkinson's disease: a randomised, double-blind, placebo-controlled trial. Lancet. 2017 Oct 7;390(10103):1664-1675. doi: 10.1016/S0140-6736(17)31585-4. Epub 2017 Aug 3. PMID 28781108
- [Background] Aviles-Olmos I, Dickson J, Kefalopoulou Z, Djamshidian A, Ell P, Soderlund T, Whitton P, Wyse R, Isaacs T, Lees A, Limousin P, Foltynie T. Exenatide and the treatment of patients with Parkinson's disease. J Clin Invest. 2013 Jun;123(6):2730-6. doi: 10.1172/JCI68295. PMID 23728174
- [Background] Chaudhuri KR, Sauerbier A, Rojo JM, Sethi K, Schapira AH, Brown RG, Antonini A, Stocchi F, Odin P, Bhattacharya K, Tsuboi Y, Abe K, Rizos A, Rodriguez-Blazquez C, Martinez-Martin P. The burden of non-motor symptoms in Parkinson's disease using a self-completed non-motor questionnaire: a simple grading system. Parkinsonism Relat Disord. 2015 Mar;21(3):287-91. doi: 10.1016/j.parkreldis.2014.12.031. Epub 2015 Jan 5. PMID 25616694
- [Background] Chou KL, Amick MM, Brandt J, Camicioli R, Frei K, Gitelman D, Goldman J, Growdon J, Hurtig HI, Levin B, Litvan I, Marsh L, Simuni T, Troster AI, Uc EY; Parkinson Study Group Cognitive/Psychiatric Working Group. A recommended scale for cognitive screening in clinical trials of Parkinson's disease. Mov Disord. 2010 Nov 15;25(15):2501-7. doi: 10.1002/mds.23362. PMID 20878991
- [Background] Hoops S, Nazem S, Siderowf AD, Duda JE, Xie SX, Stern MB, Weintraub D. Validity of the MoCA and MMSE in the detection of MCI and dementia in Parkinson disease. Neurology. 2009 Nov 24;73(21):1738-45. doi: 10.1212/WNL.0b013e3181c34b47. PMID 19933974
- [Background] Schrag A, Barone P, Brown RG, Leentjens AF, McDonald WM, Starkstein S, Weintraub D, Poewe W, Rascol O, Sampaio C, Stebbins GT, Goetz CG. Depression rating scales in Parkinson's disease: critique and recommendations. Mov Disord. 2007 Jun 15;22(8):1077-92. doi: 10.1002/mds.21333. PMID 17394234
- [Background] Peto V, Jenkinson C, Fitzpatrick R, Greenhall R. The development and validation of a short measure of functioning and well being for individuals with Parkinson's disease. Qual Life Res. 1995 Jun;4(3):241-8. doi: 10.1007/BF02260863. PMID 7613534
- [Background] Blauwendraat C, Faghri F, Pihlstrom L, Geiger JT, Elbaz A, Lesage S, Corvol JC, May P, Nicolas A, Abramzon Y, Murphy NA, Gibbs JR, Ryten M, Ferrari R, Bras J, Guerreiro R, Williams J, Sims R, Lubbe S, Hernandez DG, Mok KY, Robak L, Campbell RH, Rogaeva E, Traynor BJ, Chia R, Chung SJ; International Parkinson's Disease Genomics Consortium (IPDGC), COURAGE-PD Consortium; Hardy JA, Brice A, Wood NW, Houlden H, Shulman JM, Morris HR, Gasser T, Kruger R, Heutink P, Sharma M, Simon-Sanchez J, Nalls MA, Singleton AB, Scholz SW. NeuroChip, an updated version of the NeuroX genotyping platform to rapidly screen for variants associated with neurological diseases. Neurobiol Aging. 2017 Sep;57:247.e9-247.e13. doi: 10.1016/j.neurobiolaging.2017.05.009. Epub 2017 May 17. PMID 28602509
- [Derived] Payne T, Sassani M, Buckley E, Moll S, Anton A, Appleby M, Maru S, Taylor R, McNeill A, Hoggard N, Mazza C, Wilkinson ID, Jenkins T, Foltynie T, Bandmann O. Ursodeoxycholic acid as a novel disease-modifying treatment for Parkinson's disease: protocol for a two-centre, randomised, double-blind, placebo-controlled trial, The 'UP' study. BMJ Open. 2020 Aug 5;10(8):e038911. doi: 10.1136/bmjopen-2020-038911. PMID 32759251